CLINICAL TRIAL: NCT04509440
Title: Efficacy of Neural Prolotherapy Versus Local Corticosteroid Soft Tissue Injection for Treatment of Anserine Bursitis
Brief Title: Efficacy of Neural Prolotherapy for Treatment of Anserine Bursitis "NPCAB"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Emmanuel Kamal Aziz Saba, Principal Investigator, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0303902
Record Dates: First submitted 2020-08-04; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Anserine Bursitis
Keywords: Anserine bursitis; Neural prolotherapy; Perineural injection
MeSH Terms: interventions — Water; Solutions; Adrenal Cortex Hormones; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural prolotherapy (Experimental): Neural prolotherapy using isotonic dextrose 5% in water solution (about 3 ml). The injection was done using Lyftgot technique. The subcutaneous injections were done at sensory nerves fascial penetration points and tender areas around the anserine bursa anatomical region.
  Interventions: Drug: isotonic dextrose 5% in water (D5W) solution
- Corticosteroid group (Active Comparator): Corticosteroid with local anaesthetics (40 mg of triamcinolone acetonide (40 mg/ml) with 1.5 ml mepivacaine HCl 3% ) (local anesthetic). They were given as a single local soft tissue injection at the point of maximal tenderness on the lower medial aspect of the knee region.
  Interventions: Drug: corticosteroid with local anaesthetics (40 mg of triamcinolone acetonide (40 mg/ml) with 1.5 ml mepivacaine HCl 3% )

INTERVENTIONS:
Drug: isotonic dextrose 5% in water (D5W) solution — Neurol prolotherapy (NP) is the subcutaneous perineural injection of isotonic dextrose 5% in water (D5W) solution.
  Other Names: Subcutaneous nerual prolotherapy
  Arms: Neural prolotherapy
Drug: corticosteroid with local anaesthetics (40 mg of triamcinolone acetonide (40 mg/ml) with 1.5 ml mepivacaine HCl 3% ) — Corticosteroid with local anaesthetics (40 mg of triamcinolone acetonide (40 mg/ml) with 1.5 ml mepivacaine HCl 3% ) (local anesthetic). They were given as a single local soft tissue injection at the point of maximal tenderness on the lower medial aspect of the knee region.
  Arms: Corticosteroid group

SUMMARY:
Anserine bursitis is a common etiology of medial knee pain. It could be severe enough to limit the patient's functional abilities with affection of the quality of life. The etiology of AB is unknown. It could be bursitis, tendinitis or other unknown etiology.

The treatment of AB includes conservative and surgical treatment. Conservative treatment consists of non-pharmacologic treatment and pharmacologic treatment. Local corticosteroid injection is a treatment for refractory chronic anserine bursitis.

Neural prolotherapy is the subcutaneous perineural injection of isotonic dextrose 5% in water solution at the fascial penetration point of the sensory nerve where it reaches the subcutaneous plane and along its course. It can be used for the treatment of chronic anserine bursitis.

This study aimed to determine the efficacy of neural prolotherapy subcutaneous perineural injection versus corticosteroid local soft tissue injection therapy for relieving pain and improvement of function among patients with chronic anserine bursitis.

DETAILED DESCRIPTION:
Anserine bursitis is a common etiology of medial knee pain. It could be severe enough to limit the patient's functional abilities with affection of the quality of life. The etiology of AB is unknown. It could be bursitis, tendinitis or other unknown etiology.

The treatment of AB includes conservative and surgical treatment. Conservative treatment consists of non-pharmacologic treatment and pharmacologic treatment. Their aim is pain relieve, with subsequent improvement of function and quality of life. The non-pharmacologic treatment consisted of activity modification with avoidance of precipitating activities and physiotherapy. The pharmacologic treatment consists of non-steroidal anti-inflammatory drugs, analgesics whether oral as acetaminophen or topical preparations; or local soft tissue injection of corticosteroid. Surgical treatment is indicated after failure of conservative treatment in chronic severe and resistant cases only.

Local corticosteroid injection is a treatment for refractory chronic anserine bursitis. The mechanism of action of corticosteroid is the suppression of the inflammatory process associated with anserine bursitis. Subsequently, improvement of anserine bursitis takes place.

Neural prolotherapy is the subcutaneous perineural injection of isotonic dextrose 5% in water solution at the fascial penetration point of the sensory nerve where it reaches the subcutaneous plane and along its course. It can be used for the treatment of chronic anserine bursitis.

The mechanism of action of neural prolotherapy in anserine bursitis could be due to stimulation the release of a group of growth factors that enhance soft tissue healing in response to isotonic dextrose 5% in water solution injection. Subcutaneous injection of isotonic dextrose 5% in water solution was found to stimulate human cells to start proliferation, increase in cell protein and DNA synthesis. It stimulates the release of a group of growth factors as transforming growth factor-β and other growth factors. Another mechanism of neural prolotherapy is the treatment of neurogenic inflammation.

This study aimed to determine the efficacy of neural prolotherapy subcutaneous perineural injection versus corticosteroid local soft tissue injection therapy for relieving pain and improvement of function among patients with chronic anserine bursitis.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic anserine bursitis was based on clinical manifestations, which was the presence of pain in the medial and inferior aspect of the knee. It was increased during going upstairs and downstairs associated with tenderness on the inferomedial aspect of the knee joint about 5 cm below the medial knee joint line and occasionally local swelling. It could be associated with morning pain and stiffness.
2. Patients who were refractory to conservative treatment for at least 3 months were considered to have chronic anserine bursitis. Each knee was assessed separately for eligibility.

Exclusion Criteria:

* Symptomatic knee osteoarthritis.
* Internal derangement of the knee.
* Previous knee surgery.
* Prior surgery in the affected knee region.
* Systemic rheumatologic disorders.
* Fibromyalgia.
* Diabetes mellitus.
* Endocrine disorders.
* Metabolic disorders.
* Coagulopathy.
* Anticoagulant treatment.
* Current skin or soft tissue infection at or near the site of injection.
* Prior local soft tissue injection of corticosteroid for anserine bursitis in the past year.
* Prior neural prolotherapy for anserine bursitis in the past year.
* Patients presented with a systemic active inflammatory condition or infection.
* Pregnancy.
* Unwillingness to participate in the study.
* History of allergy to the used corticosteroid and/or local anaesthetic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMasters Universities osteoarthritis index (WOMAC) | 4 weeks
  It is a questionnaire that assesses knee pain, stiffness and physical function. The scale of difficulty for different questions was classified based on the following scale: 0=none, 1=slight, 2=moderate, 3=severe and 4=extreme). WOMAC total score ranges from 0 to 104 points. The lower scores indicate better status
assessment of overall Anserine bursitis pain severity was done using visual analogue scale | 4 weeks
  It is a visual analogue scale (VAS) (a 10-cm horizontal scale) in which it ranged from 0 (no pain), to 10 (severe intolerable pain)
patient's global assessment of AB severity was done using VAS | 4 weeks
  patient's global assessment of Anserine bursitis severity was done using VAS (a 10-cm horizontal scale) in which it ranged from 0 (negligible severity), to 10 (very severe disorder).
tenderness on the anserine bursa region | 4 weeks
  clinical assessment for the presence of tenderness on the anserine bursa region was done.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel K Saba, MD, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt